CLINICAL TRIAL: NCT03010813
Title: A Novel Robotic System for Single Port and Natural Orifice Transluminal Endoscopic Surgery: A Prospective, Single Center, Multispecialty Study
Brief Title: A Novel Robotic System for Single Port and Natural Orifice Transluminal Endoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor of Surgery, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC Ref. No.: 2016.348
Record Dates: First submitted 2016-12-24; First posted 2017-01-05 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Neoplasms; Urologic Neoplasms; Urologic Diseases; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Oral Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; ENT Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Urologic Neoplasms; Urologic Diseases; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Mouth Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Otorhinolaryngologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Novel single port robotic system (Experimental): A single port innovation designed to deliver an articulating 3D high definition camera and three fully articulating instruments through a single 25-mm cannula
  Interventions: Procedure: Robotic single port surgery and NOTES

INTERVENTIONS:
Procedure: Robotic single port surgery and NOTES — Robotic single port colorectal surgery; Robotic transanal surgery; Robotic single port urologic surgery; Transoral robotic surgery

SUMMARY:
This is a prospective, single center, multispecialty study that aimed to evaluate the clinical feasibility and safety of single port surgery and NOTES (mainly transanal and transoral surgery) using a novel single port robotic system.

DETAILED DESCRIPTION:
Background: Single port surgery and natural orifice transluminal endoscopic surgery (NOTES) are emerging minimally invasive surgery techniques which can further reduce patient trauma and enhance recovery. However, the wider adoption of these techniques is hampered by the limitation of instrumentation and technical difficulties. Robotic assistance may improve surgical capabilities during single port surgery and NOTES by providing augmented motion precision and manipulation dexterity.

Objectives: To evaluate the clinical feasibility and safety of single port surgery and NOTES (mainly transanal and transoral surgery) using a novel single port robotic system.

Design: Prospective, single center, multispecialty study consistent with a stage 1 (Innovation) study described in the Innovation, Development, Exploration, Assessment, Long-term Study (IDEAL) framework.

Subjects: Sixty consecutive patients with various benign/malignant pathologies indicated for single port colorectal/urologic surgery or transanal/transoral surgery who fulfilled all the inclusion and exclusion criteria will be recruited.

Intervention: Single port surgery and transanal/transoral surgery will be performed using the novel single port robotic system.

Study Endpoints: Primary: conversion rate and perioperative complications. Secondary: operative time, blood loss, pain scores, analgesic requirement, and length of stay.

Hypothesis: The prospective study will provide important information on the feasibility, safety, and effectiveness of the novel single port robotic system in performing single port surgery and NOTES in various surgical specialties. A positive study will provide supporting evidence for continuing development of this new technology.

ELIGIBILITY:
GENERAL INCLUSION CRITERIA FOR ALL PROCEDURES

1. Body mass index <35 kg/m2
2. Suitable for minimally invasive surgery
3. Willingness to participate as demonstrated by giving informed consent

GENERAL EXCLUSION CRITERIA FOR ALL PROCEDURES

1. Contraindication to general anesthesia
2. Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic intervention
3. Untreated active infection
4. Noncorrectable coagulopathy
5. Presence of another malignancy or distant metastasis
6. Emergency surgery
7. Vulnerable population (e.g. mentally disabled, pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Conversion rate | Up to 1 month
  An emergent change in the treatment plan to conventional minimally invasive (laparoscopic/endoscopic) surgery (i.e. the use of more than one additional port), multiport robotic surgery, or to open surgery
Perioperative complications | Up to 1 month
  Complications including intraoperative complications and all complications occurring during the hospital stay or within 30 days after discharge will be graded according to the Clavien-Dindo classification

SECONDARY OUTCOMES:
Operative time | Intraoperative
Estimated blood loss | Up to 1 month
Pain scores on a visual analog scale | Up to 1 month
Analgesic requirement | Up to 1 month
Length of hospital stay | Up to 1 month
Completeness of resection | Up to 1 month
  Pathologic examination of the resected specimen for completeness of resection
Resection margins | Up to 1 month
  Pathologic examination of the resected specimen for resection margins positivity
Number of lymph nodes harvested | Up to 1 month
  Pathologic examination of the resected specimen (malignant cases)
Anal continence after transanal surgery | Up to 1 year
  After transanal surgery; using the Cleveland Clinic Incontinence Score (Wexner's Score)
Fecal incontinence quality of life after transanal surgery | Up to 1 year
  After transanal surgery; using the validated Chinese version of the Fecal Incontinence Quality of Life Scale (FIQL)
Urinary continence after radical prostatectomy | Up to 1 year
  After radical prostatectomy; assessed by recording the number of pads used per day
Male sexual function after radical prostatectomy | Up to 1 year
  After radical prostatectomy; using the abridged version of the International Index of Erectile Dysfunction - erectile function domain score (IIEF-EF)
Renal function after nephrectomy | Up to 1 year
  After nephrectomy; using renal function blood tests for urea and creatinine
Swallowing function after transoral robotic surgery (TORS) | Up to 1 year
  After TORS; using the MD Anderson Dysphagia Inventory
Voice function after TORS | Up to 1 year
  After TORS; using the Voice Handicap Index (VHI) 30

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holsinger FC, Magnuson JS, Weinstein GS, Chan JYK, Starmer HM, Tsang RKY, Wong EWY, Rassekh CH, Bedi N, Hong SSY, Orosco R, O'Malley BW Jr, Moore EJ. A Next-Generation Single-Port Robotic Surgical System for Transoral Robotic Surgery: Results From Prospective Nonrandomized Clinical Trials. JAMA Otolaryngol Head Neck Surg. 2019 Nov 1;145(11):1027-1034. doi: 10.1001/jamaoto.2019.2654. PMID 31536129
- [Derived] Chan JYK, Tsang RK, Holsinger FC, Tong MCF, Ng CWK, Chiu PWY, Ng SSM, Wong EWY. Prospective clinical trial to evaluate safety and feasibility of using a single port flexible robotic system for transoral head and neck surgery. Oral Oncol. 2019 Jul;94:101-105. doi: 10.1016/j.oraloncology.2019.05.018. Epub 2019 May 28. PMID 31178203